CLINICAL TRIAL: NCT03253419
Title: Exploration of Home Safety Application Impact on Perceived Risk of Falling and Actual Falls Post Hospital Discharge
Brief Title: HotShOT: Home Safety Occupational Therapy
Acronym: HotShOT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in staffing and not able to do study
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Home for Life Design (Unknown)
Responsible Party: Principal Investigator, Pamela Roberts, Director and Professor, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro48620
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Hip Replacement
Keywords: Falls; Hip Replacement; Home Safety
MeSH Terms: interventions — Home Care Services

STUDY DESIGN:
Intervention Model Description: To evaluate the use of the Home for Life mobile application to examine home safety and perceived fall risk and actual falls within 2 weeks of hospital discharge for participants who have undergone hip replacement surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home Safety Application (Other): Use of Home Safety application as part of assessment for home safety. The only intervention is the use of the home safety application and identification of home safety issues by the patient using this application.
  Interventions: Other: Home for Life mobile application

INTERVENTIONS:
Other: Home for Life mobile application — Utilize home application to provide the participant with an understanding and recommendations to potentially decrease home hazards that may lead to risk of falls in their home.

SUMMARY:
The purpose of this research study is to examine home safety and fall risk for patients who have undergone hip replacement surgery. The investigators want to know whether evaluating home safety impacts perceived and real risk of falls at home. The study will utilize a fall risk assessment which is a questionnaire that focuses on perceived and real risk of falls at home, as well as a home safety assessment application, the Home for Life App. The participant will be asked about the home environment, including areas of the home such as the entrance, bedroom, and bathroom, and modification recommendations will be made to potentially increase safety.

DETAILED DESCRIPTION:
According to the Centers for Disease Control (CDC), 2.8 million older adults were treated in the emergency department for fall related injuries. Most falls are caused by a combination of risk factors, with more risk factors leading to an increased risk for falling.

People undergoing a total hip replacement can be seen as having an increased risk of falling. Once an individual discharges home from the hospital, it is during this continued post-operative period where pain and weakness continues to effect their walking ability. Additionally, if the patient has a history of falling, has a fear of falling, has visual deficits, and/or neuropathy, risk of falling increases.

Evaluating a patient's fear of falling and educating patient's regarding home safety may lead to a patient feeling increased confidence when completing daily activities with increased safety awareness.

The purpose of this study is to evaluate the use of the Home for Life mobile application to examine home safety and fall risk for patients who have undergone hip replacement surgery and are being discharged to their home.

Study Aims:

1. The first aim of this study is to assess whether completion of a home safety assessment within an acute care setting will facilitate carryover and reduce a person's actual and perceived risk of falling. The Home Safety Assessment tool will be used to make adaptation recommendations to a person's home setting based on their real and perceived risk of falling in different rooms within the home (entrance, bedroom, bathroom at a minimum). A home safety assessment is a standard in the clinical care provided by occupational therapist (OT). The use of the home safety application being an alternative method of gathering the information is for research purposes in this study and is not currently used in daily operations. During the initial evaluation, the occupational therapist will bring a tablet into the room. The tablet will have the downloaded user-friendly application. The therapist will guide the client through the components of the application, identifying different rooms in their home and asking questions pertaining to their real and perceived risk of falling within these rooms. Information obtained during this process will then be stored on RedCap.
2. The second aim of this study will be to determine if recommended adaptations in home safety impacted perceived risk of falling.
3. The third aim of this study will be to determine if the patient had a fall within two weeks post discharge.

ELIGIBILITY:
Inclusion Criteria:

* Elective total hip arthroplasty
* Discharge destination from acute care hospital is to home
* ≥ 65 years old
* Prior to admission, independent in activities of daily living

Exclusion Criteria:

* Hip replacement due to trauma
* Discharge plan to skilled nursing facility, long term care hospital or inpatient rehabilitation facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Relationship of Use of Home safety assessment and Perceived Risk of Falling | Identified during Initial evaluation
  Number of participants who identified perceived risk of falling and number of participants who used of home safety application

SECONDARY OUTCOMES:
Actual Fall and Use of application/adaptations | 2 weeks of hospital discharge
  Relationship of participant actual fall within 2 weeks of hospital discharge and use of home safety application/adaptations. Number of participants who utilized home safety application/adaptation and number of participants who had an actual fall

CONTACTS AND LOCATIONS:
Overall Officials: Richard Riggs, MD, Study Chair — Cedars-Sinai
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD at this time